CLINICAL TRIAL: NCT00438698
Title: Effect of Low Glycemic Index Diets on Glucose Control in Non-Insulin Dependent Diabetics
Brief Title: Low Glycemic Index Diets vs. High Cereal Fibre Diets in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, David Jenkins, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 04-021; CIHR RCT#: 67894 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes; Cardiovascular Disease
Keywords: Nutrition; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Glycemic Index Diet (Experimental): Diet with low glycemic index carbohydrates
  Interventions: Other: Low Glycemic Index diet
- High Fiber Diet (Active Comparator): Diet with high cereal fibre choices
  Interventions: Other: High Cereal Fibre Diets

INTERVENTIONS:
Other: Low Glycemic Index diet — Diet to emphasize carbohydrate foods low in glycemic index
  Arms: Low Glycemic Index Diet
Other: High Cereal Fibre Diets — Diet to emphasize whole wheat carbohydrate cgoices
  Arms: High Fiber Diet

SUMMARY:
Large observational studies have shown cereal fiber to protect from diabetes and heart disease. Despite the success of acarbose, an α-glucosidase hydrolase inhibitor, which lowers the glycemic index of foods containing starch, sucrose and maltodextrins, the use of diets containing low glycemic index foods still remains to be established. We will therefore provide otherwise healthy individuals with type 2 diabetes intensive counseling on food selection either to improve glucose control using high cereal fiber dietary strategies or low glycemic index foods. Studies will last 6 months with bloods taken for HbA1c, glucose and blood lipids. If the study shows a benefit for either or both diets then use of high fiber and/or low glycemic index foods in the diet may provide another potential way to improve glucose control and lower cholesterol levels in non-insulin dependent diabetes.

DETAILED DESCRIPTION:
Recruitment: Subjects will be recruited by placing advertisements in local newspapers and by distributing similar advertisements to the diabetes clinic and diabetes education programs.

Information Sessions: Approximately 1000 volunteers in groups of 10-30 with or without spouses will attend one of a number of evening information sessions run from the Risk Factor Modification Center at St. Michael's Hospital. During the sessions the exact nature of the study will be described and volunteers will have the opportunity to ask specific questions about the study and taste the high fiber and low glycemic index foods.

Screening: Potential subjects will then fill in and return to the investigators a detailed questionnaire concerning their medical history, medications (including vitamin, mineral and nutritional supplements) smoking habits, alcohol intake and exercise pattern and whether they are currently on a specific diet. Details will also be obtained concerning planned vacations. Those subjects deemed potentially eligible will be asked to give a fasting blood sample at the Risk Factor Modification Center. Individuals who meet the study criteria, are invited to return again to the Center. The principles of the diabetic diet which they are already expected to be following will be reinforced, which incorporate the key elements of an NCEP Step 2 diet (total calories from fat <30%, saturated fat <7%, polyunsaturated fat <10%, dietary cholesterol <200 mg/day).

All subjects will then be randomized to one 24-week treatment in a two-treatment parallel design.

Treatments: 1) low glycemic index dietary advice (e.g. to eat intact grain cereals, pumpernickel bread, parboiled rice, cracked wheat, pasta, peas, beans and lentils) 2) high cereal fiber diet. Background diets will be the subjects' diabetic diets, modified as above, which will conform to CDA and NCEP Step 2 guidelines. Diet histories will be recorded at weeks 0, 2, 4, 8, 12, 16 and 24. These diets will be assessed for consistency by the dietitian in the subject's presence. Where necessary, modifications in diet will be made to ensure weight maintenance. Compliance will be assessed by 7 day food records.

Duration: the study will consist of four months recruitment and patient selection, during which time estimation of individual caloric requirements will be performed, and 6 months treatment period

Study Details: Fasting blood samples are obtained at day zero and weeks 2, 4, 8, 12, 16 and 24 of each study period. Twenty-four hour urine for urinary C-peptide analyses will be obtained immediately prior to the beginning of the study and at the end of each 24-week treatment phase.

Palatability and satiety: subjects will record their ratings using a 9-point bipolar semantic scale at weekly intervals during each study phase.

Anthropometric measures: height at recruitment, waist and hip circumference, and body composition will be taken immediately prior to and at the end of each study phase. Body weight and blood pressure will be measured at clinic visits.

This study will help to indicate whether dietary advice can make a significant difference to glycemic control as has been the case with drug therapy to reduce postprandial glycemia.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women with type 2 diabetes treated with diet plus oral hypoglycemic agents (Sulfonylureas, Biguanides, Thiazolidinediones , and new secretagogues (Repaglinide)) at a stable dose for at least 3 months prior to starting the study
* HbA1c between 6.5 and 8.0% at recruitment
* living within a 40 km radius of St. Michael's Hospital
* Diabetes diagnosed > 6 months prior to randomization

Exclusion Criteria:

* diabetic complications: clinically significant gastroparesis, retinopathy, nephropathy, neuropathy, hepatic disease, or CHD (current clinically significant CHD e.g. unstable angina)
* taking insulin or acarbose
* smoking or significant alcohol intake (> 1 drink/day)
* serum triglycerides > 4.0 mmol/L

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2004-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | 6 months
Change in Fasting Glucose | 6 months

SECONDARY OUTCOMES:
serum FFA | 6 months
C-peptide | 6 months
CRP | 6 months
IGF-I | 6 months
IGFBP-3 | 6 months
Serum apo AI | 6 months
apo B | 6 months
apo Lp(a) | 6 months
amino acids | 6 months
Plasma lipids and lipoproteins (TG, LDL, HDL) | 6 months
Oxidized LDL | 6 months
Change in Urinary creatinine | 6 months
urea | 6 months
Urinary C-peptide | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, MD, PhD, Principal Investigator — University of Toronto, St. Michael's Hospital; Cyril WC Kendall, PhD, Study Director — University of Toronto, St. Michael's Hospital
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kavanagh ME, Back S, Chen V, Glenn AJ, Viscardi G, Houshialsadat Z, Sievenpiper JL, Kendall CWC, Jenkins DJA, Chiavaroli L. The Portfolio Diet and HbA1c in Adults Living with Type 2 Diabetes Mellitus: A Patient-Level Pooled Analysis of Two Randomized Dietary Trials. Nutrients. 2024 Aug 23;16(17):2817. doi: 10.3390/nu16172817. PMID 39275135
- [Derived] Ha V, Viguiliouk E, Kendall CWC, Balachandran B, Jenkins DJA, Kavsak PA, Sievenpiper JL. Effect of a low glycemic index diet versus a high-cereal fibre diet on markers of subclinical cardiac injury in healthy individuals with type 2 diabetes mellitus: An exploratory analysis of a randomized dietary trial. Clin Biochem. 2017 Dec;50(18):1104-1109. doi: 10.1016/j.clinbiochem.2017.09.021. Epub 2017 Sep 25. PMID 28958804
- [Derived] Jenkins DJ, Srichaikul K, Kendall CW, Sievenpiper JL, Abdulnour S, Mirrahimi A, Meneses C, Nishi S, He X, Lee S, So YT, Esfahani A, Mitchell S, Parker TL, Vidgen E, Josse RG, Leiter LA. The relation of low glycaemic index fruit consumption to glycaemic control and risk factors for coronary heart disease in type 2 diabetes. Diabetologia. 2011 Feb;54(2):271-9. doi: 10.1007/s00125-010-1927-1. Epub 2010 Oct 27. PMID 20978741
- [Derived] Jenkins DJ, Kendall CW, McKeown-Eyssen G, Josse RG, Silverberg J, Booth GL, Vidgen E, Josse AR, Nguyen TH, Corrigan S, Banach MS, Ares S, Mitchell S, Emam A, Augustin LS, Parker TL, Leiter LA. Effect of a low-glycemic index or a high-cereal fiber diet on type 2 diabetes: a randomized trial. JAMA. 2008 Dec 17;300(23):2742-53. doi: 10.1001/jama.2008.808. PMID 19088352